CLINICAL TRIAL: NCT05628961
Title: An Open-Label, First-In-Human Study of Single Oral Doses of HOPO 14-1 Evaluating Safety, Tolerability, Pharmacokinetics, and Excretion in Healthy Participants
Brief Title: Study of Single Oral Doses of HOPO 14-1 Evaluating Safety, Tolerability, Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SRI International (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SRI-HOPO-01
Record Dates: First submitted 2022-11-17; First posted 2022-11-29 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Toxicity;Chemical
Keywords: Internal Radionuclide Contamination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1: 100 mg (Experimental): Participants receive an oral single dose of HOPO 14-1 in the fasted condition on Day 1.
  Interventions: Drug: HOPO 14-1
- Cohort 2: 200 mg (Experimental): Participants receive an oral single dose of HOPO 14-1 in the fasted condition on Day 1.
  Interventions: Drug: HOPO 14-1
- Cohort 3: 500 mg (Experimental): Participants receive an oral single dose of HOPO 14-1 in the fasted condition on Day 1.
  Interventions: Drug: HOPO 14-1
- Cohort 4: 1200 mg (Experimental): Participants receive an oral single dose of HOPO 14-1 in the fasted condition on Day 1.
  Interventions: Drug: HOPO 14-1
- Cohort 5: 2500 mg (Experimental): Participants receive an oral single dose of HOPO 14-1 in the fasted condition on Day 1.
  Interventions: Drug: HOPO 14-1
- Cohort 6: 5000 mg (Experimental): Participants receive an oral single dose of HOPO 14-1 in the fasted condition on Day 1.
  Interventions: Drug: HOPO 14-1
- Cohort 7: 7500 mg (Experimental): Participants receive an oral single dose of HOPO 14-1 in the fasted condition on Day 1.
  Interventions: Drug: HOPO 14-1

INTERVENTIONS:
Drug: HOPO 14-1 — HOPO 14-1 contains the active pharmaceutical ingredient (API) 3, 4, 3-LI(1, 2-HOPO) formulated with a permeability enhancer, sodium oleate, in capsule form.

SUMMARY:
The study objectives are to define the safety and tolerability profile of oral, single ascending dose (SAD) levels of HOPO 14-1 capsules in cohorts of healthy participants and to assess the pharmacokinetic (PK) and excretion profile of HOPO 14-1. The study hypothesis is that a single dose of HOPO 14-1 will be safe and tolerable up to 7500 mg.

DETAILED DESCRIPTION:
The currently available therapy for radionuclide internal contamination is suboptimal. Pharmacological and toxicological data support the clinical development of HOPO 14-1 for decorporation of radionuclides.

ELIGIBILITY:
Inclusion Criteria:

* Ability of participant to understand the requirements of the study, provide written informed consent, and agree to abide by the study requirements
* Agree to use contraception from time of screening until 14 days after dosing (Day 14) if female is of childbearing potential or male is with female partner of childbearing potential.
* In good general health based on medical history, physical examination (PE), and screening evaluations.
* Negative urine screen for drugs of abuse (except if participant provides prescription justifying use prior to urine screen).
* Body weight ≥ 50 kilogram (kg) and ≤ 110 kg. If body weight is over 110 kg, then body mass index (BMI) will be considered and must be ≤ 40 kg/m^2.

Exclusion Criteria:

* Inability or unwillingness of a participant to give written informed consent or comply with study protocol.
* Any hematology, chemistry, coagulation, or urinalysis value on screening labs defined in the United States Food and Drug Administration (FDA) Guidance for Industry Toxicity Grading Scale as Grade 1 or higher.
* Any clinically significant electrocardiogram (ECG) abnormality
* Pregnant or breastfeeding
* Active substance abuse or history of any medical or psychiatric condition that would jeopardize the participant's safety or the participant's ability to comply with the protocol.
* Received an organ transplant (solid or bone marrow).
* Received a blood transfusion within 3 months of dosing.
* Difficulty swallowing tablets or capsules.
* Febrile illness or significant infection within 7 days of dosing.
* Symptoms of hypotension (lightheadedness, syncope, balance disturbances, or extreme fatigue) within 48 hours of dosing.
* Hepatitis B virus surface antigen (HBsAg) positive or serologic (antibody positive) evidence of infection with hepatitis C virus (HCV) or human immunodeficiency virus (HIV).
* Tested positive for SARS-CoV-2 (COVID-19) within 21 days of dosing.
* Chelation therapy (e.g., ethylenediaminetetraacetic acid [EDTA], diethylenetriamine pentaacetate [DTPA]) in the past year.
* Use of laxatives, antibiotics, and/or antacids within 7 days of dosing.
* Use of investigational drugs within 60 days of dosing or 5 half-lives, whichever is longer.
* Received a vaccination within 30 days of dosing.
* Potential allergic reaction to product (oleic acid or HOPO 14-1 product).
* Past or current medical problems or findings from physical examination (PE) or laboratory testing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Adverse Events | Up to 14 days
Number of Participants with One or More Drug-Related Adverse Events | Up to 14 days
Number of Participants with One or More Adverse Events by Maximum Severity | Up to 14 days
Number of Participants with One or More Serious Adverse Events | Up to 14 days

SECONDARY OUTCOMES:
Observed Maximum Plasma Concentration (Cmax) | Up to Day 7
Observed Time to Reach Cmax (Tmax) | Up to Day 7
Area Under the Plasma Concentration Time Curve up to the Last Blood Collection Time with a Measurable Concentration (AUClast) | Up to Day 7
Extrapolated to Infinity (AUC0-inf) | Up to Day 7
Terminal Half-Life (t 1/2) | Up to Day 7
Apparent Volume of Distribution after Oral Administration (V/F) | Up to Day 7
Oral Systemic Clearance Rate (CL/F) | Up to Day 7
Cumulative Amount Excreted in Urine | Up to Day 7
Cumulative Amount Excreted in Feces | Up to Day 7

CONTACTS AND LOCATIONS:
Locations (1):
- SRI International Clinical Trials Unit, Plymouth, Michigan, United States